CLINICAL TRIAL: NCT04848389
Title: Optimization of the Nursing Time After the Use of Tissue Adhesives During the Chest Port Placement on Patients Treated With Chemotherapy, a Randomized Trial Versus Sutures
Brief Title: Optimization of the Nursing Time After the Use of Tissue Adhesives During the Chest Port Placement on Patients Treated With Chemotherapy Versus Sutures
Acronym: PAC_COLLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAC_COLLE
Record Dates: First submitted 2021-03-23; First posted 2021-04-19 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin adhesive (Experimental): The scar is closed in 2 planes. The subcutaneous plane is closed with an absorbable 3/0 vicryl-type thread, the cutaneous plane is closed by applying skin adhesive. A drying time of 25 seconds is necessary to obtain a satisfactory seal.
  Interventions: Procedure: Skin Adhesive procedure
- Standard suture (Other): The scar is closed in 2 planes. The subcutaneous plane is closed with an absorbable 3/0 vicryl-type thread, the cutaneous plane is closed with the same thread with a subcutaneous stitch.
  Interventions: Procedure: Standard suture procedure

INTERVENTIONS:
Procedure: Skin Adhesive procedure — The scar is closed in 2 planes. The subcutaneous plane is closed with an absorbable 3/0 vicryl-type thread, the cutaneous plane is closed by applying skin adhesive. A drying time of 25 seconds is necessary to obtain a satisfactory seal.
  Arms: Skin adhesive
Procedure: Standard suture procedure — The scar is closed in 2 planes. The subcutaneous plane is closed with an absorbable thread of the 3/0 Vicryl-type, the cutaneous plane is closed with the same thread with an subcutaneous stitch.
  Arms: Standard suture

SUMMARY:
Skin adhesive (Octyl cyanoacrylate - LIQUID BAND©) is increasingly used instead of suture for sutures on the superficial plane of the skin.

It is frequently used in children, in traumatology and in plastic surgery. Several randomized trials have shown satisfactory results of the glue compared to suture in terms of infections and scar dehiscence, and aesthetics after abdominoplasty and mammoplasty.

In the field of port-a-cath® placement in oncology:

* The use of skin adhesive can save substantial nursing time, which makes it possible to consider the transition of this technique into routine patient management. Potential benefits include nurses managing large numbers of patients in day hospitals, and patients no longer needing a nurse for suture removal.
* Cancer and chemotherapy toxicity can alter patients' body image and view of themselves. The presence of a scar can be traumatic for some patients. The second goal of this study is to test whether the use of glue can improve the appearance of the scar following port-a-cath® placement, an area in which there are divergent results.

ELIGIBILITY:
Inclusion Criteria:

* Patient with age ≥ 18 years
* Patient followed in day hospitalization in Oncology
* Patient requiring a first CP for chemotherapy
* Patient affiliated to a healthcare system
* French-speaking patient
* Patient who has given his free, informed and express oral consent

Exclusion Criteria:

* Patient followed in the Pneumology department
* Patient treated outside the GHPSJ
* Patient with a CP for another indication than chemotherapy (nutrition, antibiotic therapy)
* Patients with comprehension problems
* Patients with behavior issues
* Pregnant women
* Patients under guardianship or curatorship
* Patients deprived of liberty
* Patients under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
The tissue adhesive, a technique adapted to save the nursing time. (Timed nursing time for PAC infusion) | 1 month
  This outcome corresponds to the Timed nursing time for PAC infusion in the first cycle of chemotherapy and comparison between the 2 arms.

SECONDARY OUTCOMES:
Physical shape of the scar (POSAS scale) | 1 month
  This outcome correspond to the POSAS scale which is a reliable and valid scar assessment scale that measures scar quality from two perspectives: the patient and the clinician. The POSAS measures scar quality in all types of scars. The observer scale of the POSAS consists of six items (vascularity, pigmentation, thickness, relief, pliability and surface area). All items are scored on a scale ranging from 1 ('like normal skin') to 10 ('worst scar imaginable'). The sum of the six items results in a total score of the POSAS observer scale. Categories boxes are added for each item. Furthermore, an overall opinion is scored on a scale ranging from 1 to 10. All parameters should preferably be compared to normal skin on a comparable anatomic location.
Patient's comfort | 30 days
  This outcome correspond to the assessment of the patient's comfort at D30 during the implantation with the tissue adhesive comparing to the sutures.1. In the time between the installation of PAC and visit , did patient use for PAC? a home health aide or a nurse? 2. Did patient visit his general practitioner in this interval for your PAC? Yes or No 3. On a scale of 0 to 10, what pain are patient experiencing today? 4. On a scale of 0 to 10, how much discomfort are patient experiencing today? 5. Following PACplacement, how soon were patient able to resume showering in days? 6. Following the placement of the PAC, how soon were patient able to resume a normal life in days?

CONTACTS AND LOCATIONS:
Overall Officials: Lynda SALMI, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, Groupe Hospitalier Paris Saint-Joseph, France

REFERENCES:
- [Background] Vida VL, Barzon E, Sabiu C, De Franceschi M, Padalino MA, Stellin G. The use of "2-octyl cyanoacrylate" as skin adhesive in pediatric and congenital cardiac surgery. Minerva Pediatr. 2015 Apr;67(2):111-6. Epub 2015 Jan 21. PMID 25604588
- [Background] Parvizi D, Friedl H, Schintler MV, Rappl T, Laback C, Wiedner M, Vasiljeva A, Kamolz LP, Spendel S. Use of 2-octyl cyanoacrylate together with a self-adhering mesh (Dermabond Prineo) for skin closure following abdominoplasty: an open, prospective, controlled, randomized, clinical study. Aesthetic Plast Surg. 2013 Jun;37(3):529-37. doi: 10.1007/s00266-013-0123-3. Epub 2013 Apr 24. PMID 23613192
- [Background] Nipshagen MD, Hage JJ, Beekman WH. Use of 2-octyl-cyanoacrylate skin adhesive (Dermabond) for wound closure following reduction mammaplasty: a prospective, randomized intervention study. Plast Reconstr Surg. 2008 Jul;122(1):10-18. doi: 10.1097/PRS.0b013e318171524b. PMID 18594354
- [Background] Martin JG, Hollenbeck ST, Janas G, Makar RA, Pabon-Ramos WM, Suhocki PV, Miller MJ, Sopko DR, Smith TP, Kim CY. Randomized Controlled Trial of Octyl Cyanoacrylate Skin Adhesive versus Subcuticular Suture for Skin Closure after Implantable Venous Port Placement. J Vasc Interv Radiol. 2017 Jan;28(1):111-116. doi: 10.1016/j.jvir.2016.08.009. Epub 2016 Nov 9. PMID 27836404
- [Background] Singer AJ, Arora B, Dagum A, Valentine S, Hollander JE. Development and validation of a novel scar evaluation scale. Plast Reconstr Surg. 2007 Dec;120(7):1892-1897. doi: 10.1097/01.prs.0000287275.15511.10. PMID 18090752
- [Background] Liberale G, El Houkayem M, Viste C, Bouazza F, Moreau M, El Nakadi I, Veys I. Evaluation of the perceptions and cosmetic satisfaction of breast cancer patients undergoing totally implantable vascular access device (TIVAD) placement. Support Care Cancer. 2016 Dec;24(12):5035-5040. doi: 10.1007/s00520-016-3368-y. Epub 2016 Aug 5. PMID 27495928